CLINICAL TRIAL: NCT01842334
Title: D-cycloserine (DCS) Pretreatment + Cognitive Behavioral Therapy and Nicotine Replacement Therapy for Smoking Cessation
Brief Title: D-cycloserine (DCS) Pretreatment + CBT + Nicotine Replacement Therapy for Smoking Cessation (DCS)
Acronym: DCS
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: left institution protocol closed
Sponsor: Mclean Hospital (Other)
Collaborators: American Lung Association (Other)
Responsible Party: Principal Investigator, Kevin P. Hill, MD, MHS, Assistant Professor of Psychiatry, Mclean Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2012P001707
Record Dates: First submitted 2013-04-25; First posted 2013-04-29 (Estimated); Results first posted 2018-08-01 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Nicotine Dependence; Smoking Cessation
Keywords: Nicotine Dependence; Smoking Cessation; D-cycloserine
MeSH Terms: conditions — Tobacco Use Disorder; Smoking Cessation | interventions — Cognitive Behavioral Therapy; Nicotine Replacement Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- D-cycloserine (Experimental): 250 mg D-cycloserine once weekly an hour before receiving cognitive behavioral therapy treatment along with Nicotine Replacement Therapy.
  Interventions: Behavioral: Cognitive Behavioral Therapy; Drug: Nicotine Replacement Therapy
- Placebo (Placebo Comparator): one placebo capsule once weekly an hour before receiving cognitive behavioral therapy treatment along with Nicotine Replacement Therapy
  Interventions: Behavioral: Cognitive Behavioral Therapy; Drug: Nicotine Replacement Therapy

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — CBT administered to to both DCS and placebo group.
  Other Names: CBT
Drug: Nicotine Replacement Therapy — NRT administered to both DCS and placebo group.
  Other Names: NRT

SUMMARY:
1. Compare the relative efficacy of ten weeks of once weekly 250 mg D-cycloserine (DCS) vs. placebo (both in conjunction with cognitive behavioral therapy (CBT) and nicotine replacement therapy (NRT) on reducing cigarette smoking in treatment-seeking nicotine-dependent outpatients.
2. Compare the relative efficacy of ten weeks of once weekly 250 mg DCS vs. placebo on the process of extinction and the memory encoding process.

DETAILED DESCRIPTION:
The investigators will conduct a Stage 1 pilot feasibility study at McLean Hospital to develop a medication to treat nicotine dependence. In a randomized, double-blind, placebo-controlled trial, 40 nicotine-dependent participants ages 18-65 will receive cognitive behavioral therapy (CBT) and nicotine replacement therapy (NRT) over a 10- week period, with half receiving D-cycloserine (DCS) pretreatment and half receiving placebo. Participants will receive either 250 mg DCS or placebo prior to weekly CBT sessions in addition to NRT over a 10-week treatment period. The investigators also aim to determine the effects of DCS on performance on neuropsychological tests. A 10-week treatment period will be followed by follow-up assessments including neuropsychological tests at 1 and 3 months post-treatment. Primary outcomes will include smoking as measured by carbon monoxide levels and self-report measurements.

ELIGIBILITY:
Inclusion Criteria:

1) Age range 18-65 years; 2) DSM-IV diagnosis of nicotine dependence, based on the Structured Clinical Interview for DSM-IV (SCID) (First et al. 1996); 3) express a desire to quit cigarette smoking within the next 30 days; 4) smokes greater than or equal to 10 cigarettes per day and less than or equal to 20 cigarettes per day; 5) an expired carbon monoxide (CO) determination greater than or equal to 10 ppm over ambient values; 6) for women of childbearing age, a negative pregnancy test at screening with agreement to use adequate contraception to prevent pregnancy and multiple subsequent pregnancy tests; 7) consent for us to communicate with their prescribing clinician; 8) furnish the names of 2 locators, who would assist study staff in locating them during the study period; 9) live close enough to McLean Hospital to attend study visits; 10) plan to remain in the Boston area for the next 4 months; and 11) are willing and able to sign informed consent.

Exclusion Criteria:

1) Current diagnosis of other drug or alcohol dependence (other than nicotine); 2) significant cardiac disease; 3) current serious psychiatric illness or history of psychosis, schizophrenia, bipolar type I disorder (taking psychiatric medications, aside from wellbutrin, is not an exclusionary criterion); 4) have a current medical condition (including significant laboratory abnormalities, such as liver function tests >5 times the upper limit of normal range) that could prevent regular study attendance; 5) have mental retardation or organic mental disorder; 6) exhibit acutely dangerous or suicidal behavior; 7) are pregnant, nursing, or, if a woman of childbearing potential, not using a form of birth control judged by the Principal Investigator to be effective; 8) current NRT or other smoking cessation treatment;9) current CBT for smoking cessation; 10) current smokeless tobacco use; 11) inability to read or write in English;12) has epilepsy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin P. Hill, MD, MHS, Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 9 out of the 21 subject screened did not qualify for randomization. 6 of the subjects were no longer interested in participating after the screening visit, 2 did not return repeated phone calls by study staff and 1 subject did not qualify due to being on probation.
Period: Overall Study
Arm/Group | D-cycloserine | Placebo
Started | 5 | 7
Completed | 2 | 3
Not Completed | 3 | 4
Not completed — Withdrawal by Subject | 3 | 3
Not completed — Moved away mid-study | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | D-cycloserine | Placebo | Total
Number analyzed (Participants) | 5 | 7 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 30 (6.96) | 39.57 (15.79) | 35.58 (13.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 3 | 4 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 4 | 6 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Baseline Cigs/Day [Mean (Standard Deviation); unit: cigarettes/day] | 13.34 (2.18) | 12.87 (2.01) | 13.04 (1.97)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Cigarette Smoking in Treatment Seeking Nicotine Dependent Outpatients
Description: Cigarette smoking at 10 weeks as measured by carbon monoxide levels and self-report measurements.
Time Frame: During Week 10
Population: Only the 5 completers of this study who made it to week 10 could have this measure analyzed.
Measure: Mean (Standard Deviation); unit: Cigarettes/day
Arm/Group | D-cycloserine | Placebo
Number analyzed (Participants) | 2 | 3
Cigarettes/day | 2.57 (3.63) | 0.29 (0.25)

ADVERSE EVENTS:
Time Frame: Adverse even data was collected from the baseline visit until the end of the study (14 weeks after baseline)
Arm/Group | D-cycloserine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/7
Other Adverse Events (participants affected / at risk) | 1/5 | 0/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | D-cycloserine (N=5) | Placebo (N=7)
Nausea due to Nicotine Patch (General disorders) | 1 (1) | 0 (0) — Only 1 subject in the study reported nausea associated with the nicotine patch. The nicotine patch dosage was decreased from 21mg to 14mg by the PI following the procedure outlined in the protocol.

LIMITATIONS AND CAVEATS:
Due to lack of sufficient funds/resources, the sample size for this study is not large enough to extract any conclusive results. The high number of subjects withdrawing from the study early also hinders any possible conclusions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-09-10): https://cdn.clinicaltrials.gov/large-docs/34/NCT01842334/Prot_SAP_000.pdf